CLINICAL TRIAL: NCT02495272
Title: The Effect of the Timing of Uterotonic Administration in the Third Stage of Labour on Postpartum Hemorrhage
Brief Title: Postpartum Uterotonic Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Collaborators: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Eser Sefik Ozyurek, MD, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Kanuni-Bagcilar
Record Dates: First submitted 2015-04-09; First posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Postpartum Bleeding
Keywords: Postpartum hemorrhage; Third stage of labour; Oxytocin; Uterotonics; Active management of third stage of labour
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Oxytocin 10IU im was administered after placental delivery
  Interventions: Drug: Oxytocin
- Study Group (Experimental): Oxytocin 10IU im was administered after the anterior shoulder could be seen.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin 10IU Administered intramuscularly.
  Other Names: PostuitrinFort Amp I.E.Ulagay

SUMMARY:
The investigators are planning to determine the effect of the timing of oxytocin administration on the amount of blood loss, necessity for additional medical or surgical interventions.

DETAILED DESCRIPTION:
The investigators are studying the effects of the timing of intramuscular oxytocin administration in the third stage of labour. The investigators are measuring the postpartum blood loss: quantitatively in the postpartum 1st hour and indirectly by the decrease in the hemoglobin-haematocrit levels in the postpartum 24th hour. The investigators are monitoring the length of the third stage of labour, and the need for extra uterotonics and/or surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Cephalic presentation
* Singleton pregnancy
* Gestational age >35 weeks,
* In active labour.
* Expected fetal birth weight 2500-4500 grams.

Exclusion Criteria:

* Acute Fetal Distress
* Conversion to abdominal delivery
* Persistent high blood pressure (>140/90mmHg)
* Placenta Previa
* Ablatio placenta
* Previous C-Section
* Uterine scar
* Postpartum hemorrhage in previous pregnancies.
* Hydramnios
* Maternal infection
* Forceps/Vacuum Assisted deliveries
* Abnormal placentation ( Placenta accreta, increta or percreta)
* Coagulation Defects
* Hemoglobin < 8g/dl

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum blood loss | Participants will be followed for the duration of hospital stay, an expected average of 24 hour
  Quantitative collection of blood loss.
Postpartum blood loss >500cc | Participants will be followed for the duration of hospital stay, an expected average of 24 hour
  Number of participants whose blood loss is higher than 500cc.

SECONDARY OUTCOMES:
Need for additional uterotonics | Participants will be followed for the duration of hospital stay, an expected average of 24 hour
  Additional uterotonics (Oxytocin 10IU; Cytotec tb Rectal and/or vaginal) were administered if postpartum blood loss >500ml OR uterine atony was observed OR sudden excessive hemorrhage was encountered.
Postpartum transfusion | Participants will be followed for the duration of hospital stay, an expected average of 24 hour.
Manual removal of the placenta. | At first hour after delivery of the fetus
Duration of the third stage of labour. | Participants will be followed for the duration of labor unit stay, an expected average of one hour
Drop in the hemoglobin and hematocrit levels | At the 24th hour,postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Burak Ozkose, MD, Study Chair — Kanuni Sultan Suleyman Teaching and Research Hospital, Istanbul; Dogukan Yildirim, MD, Principal Investigator — Kanuni Sultan Suleyman Teaching and Research Hospital, Istanbul; Eser S Ozyurek, MD, Study Chair — Bagcilar Training and Research Hospital; Batuhan Ustun, MD, Study Chair — Kanuni Sultan Suleyman Teaching and Research Hospital, Istanbul
Locations (1):
- Kanuni Sultan Suleyman Teaching and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Oguz Orhan E, Dilbaz B, Aksakal SE, Altinbas S, Erkaya S. Prospective randomized trial of oxytocin administration for active management of the third stage of labor. Int J Gynaecol Obstet. 2014 Nov;127(2):175-9. doi: 10.1016/j.ijgo.2014.05.022. Epub 2014 Jul 17. PMID 25108586